CLINICAL TRIAL: NCT04349358
Title: 18F-Fluorocholine (FCH) Versus 18F-Fluorodesoxyglucose (FDG) PET/CT in Detection of Lesions in Patients With Multiple Myeloma
Brief Title: FCH vs FDG PET/CT in Detection of Lesions in Patients With Multiple Myeloma (MIM)
Acronym: MIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-003627-38
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: PET/CT; FDG; Fluorocholine (18F) FCH
MeSH Terms: conditions — Multiple Myeloma; Nuchal bleb, familial | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG and FCH PET/CT (Other)
  Interventions: Other: FDG and FCH PET/CT

INTERVENTIONS:
Other: FDG and FCH PET/CT — * during the initial myeloma check-up : FDG and FCH PET/CT exams (maximum 21 days after inclusion)
  * just before maintenance treatment, respecting a minimum interval of 2 weeks after the last course of chemotherapy : FDG and FCH PET/CT exams

SUMMARY:
Hybrid positron emission tomography/computed tomography (PET/CT) has now become available to detect tumors in patients with multiple myeloma. The radioactive glucose 18F-fluorodeoxyglucose (FDG) is the most widely used tracer but findings suggest that PET/CT reveal more lesions when using FCH.

In this study, FDG is compared with a more recent metabolic tracer, 18F-fluorocholine (FCH), for the detection of multiple myeloma lesions at time of initial extension assessment.

The principal objective of this sudy is to compare the number of suspected hypermetabolic foci of myeloma detected by 18F-fluorocholine PET and by 18F-fluorodeoxyglucose PET during the initial extension assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with initial diagnosis of multiple myeloma has just been established
* Therapeutic indication and eligible for a HSC autograft (if the HSC autograft could not be performed, the patient will still be retained in the study).
* Status ECOG 0, 1 or 2
* Age ≥ 18 and < 75 ans years
* Effective contraception for women
* Informed consent signed
* Patient able to lie flat for 30 minutes
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient diagnosed with a diagnosis of MGUS (Monoclonal Gammapathy of Undetermined Significance = monoclonal gammopathy of undetermined significance), indolent myeloma ("smoldering myeloma"), non-secreting myeloma or recurrent myeloma,
* Patient already under treatment for myeloma.
* Patient not eligible for intensive treatment followed by a HSC autograft.
* Patient with concomitant neoplasia
* Patient with a history of hematological or solid neoplasia, except if it is a basal cell carcinoma of the skin or an adenocarcinoma in situ of the uterine cervix.
* Patient with a history of sarcoidosis
* Uncontrolled diabetes.
* Patient treated with long-term corticosteroids
* Patient being treated with hematopoietic growth factors
* Patient in sepsis.
* Claustrophobic patient.
* Refusal of patient consent.
* Pregnant or lactating woman.
* Women of childbearing potential without effective contraception.
* Person deprived of liberty or under guardianship
* Impossibility to submit to the medical follow-up of the trial for geographic, social or psychological reasons.
* History of allergic reaction attributed to 18F-fluorodeoxyglucose or to 18F-fluorocholine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
number of hypermetabolic foci of myeloma detected by FCH PET versus by FDG PET during the initial extension assessment | before maintenance treatment
  PET/CT

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - CHU de Dijon, Dijon